CLINICAL TRIAL: NCT06720987
Title: A Phase 1/1b, Open-label, Multicenter, Dose Escalation and Dose Optimization Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of KQB365 as Monotherapy and in Combination With Anti-cancer Agents in Participants With Advanced Solid Malignancies With KRAS G12S or G12C Mutations
Brief Title: A Study to Investigate the Safety and Efficacy of KQB365 as Monotherapy and in Combination in Participants With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kumquat Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQB365-101
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: KRAS G12C Mutation; KRAS G12S Mutation; Solid Tumor Malignancies; CRC (Colorectal Cancer)
Keywords: cetuximab; KQB365
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Monotherapy Dose Escalation (Experimental): Drug: KQB365
  - Intravenous KQB365
  Interventions: Drug: KQB365
- Combo Therapy Dose Escalation (Experimental): Drug: KQB365 - Intravenous KQB365
  Drug:
  - Intravenous cetuximab
  Interventions: Drug: KQB365; Drug: Cetuximab
- Monotherapy Dose Expansion - RP2D (Experimental): Drug: KQB365
  - Intravenous KQB365
  Interventions: Drug: KQB365
- Monotherapy Dose Expansion - RP2D-1 (Experimental): Drug: KQB365
  - Intravenous KQB365
  Interventions: Drug: KQB365
- Combo Therapy Dose Expansion - RP2D (Experimental): Drug: KQB365 - Intravenous KQB365
  Drug:
  - Intravenous cetuximab
  Interventions: Drug: KQB365; Drug: Cetuximab
- Combo Therapy Dose Expansion - RP2D-1 (Experimental): Drug: KQB365 - Intravenous KQB365
  Drug:
  - Intravenous cetuximab
  Interventions: Drug: KQB365; Drug: Cetuximab

INTERVENTIONS:
Drug: KQB365 — Intravenous KQB365
Drug: Cetuximab — Intravenous cetuximab
  Arms: Combo Therapy Dose Escalation; Combo Therapy Dose Expansion - RP2D; Combo Therapy Dose Expansion - RP2D-1

SUMMARY:
The goal of this clinical trial is to learn if KQB365 works to treat advanced solid tumor cancer in adults. It will also learn about the safety of KQB365. The main questions it aims to answer are:

* What is the safe dose of KQB365 by itself or in combination with cetuximab?
* Does KQB365 alone or in combination with cetuximab decrease the size of the tumor?
* What happens to KQB365 in the body?

Participants will:

* Receive KQB365 infusion weekly alone or in combination with cetuximab
* Visit the clinic about 9 times in the first 6 weeks, and then once every week after that.

ELIGIBILITY:
Inclusion Criteria:

* PART 1 (monotherapy): Histologically confirmed diagnosis of a solid tumor malignancy with either a KRAS G12C or KRAS G12S mutation.
* PART 1 (combo therapy) & PART 2: Histologically confirmed diagnosis of adenocarcinoma of the colon or rectum with either a KRAS G12C or KRAS G12S mutation.
* Unresectable or metastatic disease
* No available treatment with curative intent
* Adequate organ function
* Measurable disease per RECIST v1.1

Exclusion Criteria:

* Active primary central nervous system tumors
* Cardiac abnormalities
* Active interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experience treatment-emergent adverse events, serious adverse events, and dose-limiting toxicities (Part 1) | From enrollment to the end of treatment
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of AEs, SAEs, and DLTs, from first dose of study treatment to 30 days after last dose of study treatment.
Recommended Phase 2 Dose (RP2D) (Part 1) | up to 35 months
  Evaluate safety and assess number of patients with dose-limiting toxicity to determine the RP2D.
Efficacy and Optimal Biologic Dose of study treatment, as measured by Objective Response Rate (ORR) (Part 2) | up to 35 months
  ORR is the proportion of subjects that experience confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 during the time period from 1st dose of study treatment until last dose.

SECONDARY OUTCOMES:
Concentration-time curve (AUC) | up to 35 months
Maximum plasma concentration (Cmax) | up to 35 months
Time to maximum plasma concentration (tmax) | up to 35 months
Overall survival (OS) | up to 35 months
Progression-free survival (PFS) | up to 35 months
  using RECIST v1.1
Overall response rate (ORR) | up to 35 months
  using RECIST v1.1
Duration of response (DOR) | up to 35 months
  using RECIST v1.1
Time to response (TTR) | up to 35 months
  using RECIST v1.1
Disease control rate (DCR) | up to 35 months
  using RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Mayo Clinic, Phoenix, Phoenix, Arizona
  - Sarah Cannon Cancer Institute at HealthONE, Denver, Colorado
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, LLC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No